CLINICAL TRIAL: NCT00561951
Title: A 12-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter, Dose-Finding Study To Evaluate The Efficacy, Tolerability And Safety Of Fesoterodine In Comparison To Placebo In Patients With Overactive Bladder.
Brief Title: Dose-Finding Study To Evaluate The Efficacy, Tolerability And Safety Of Fesoterodine In Comparison To Placebo For Overactive Bladder.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A0221005
Record Dates: First submitted 2007-11-19; First posted 2007-11-21 (Estimated); Results first posted 2010-09-09 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — fesoterodine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fesoterodine fumarate 4 mg (Double-Blind) (Experimental)
  Interventions: Drug: fesoterodine fumarate
- Placebo (Double-Blind) (Placebo Comparator)
  Interventions: Drug: Placebo
- Fesoterodine fumarate 8 mg (Double-Blind) (Experimental)
  Interventions: Drug: fesoterodine fumarate

INTERVENTIONS:
Drug: fesoterodine fumarate — 8mg tablets OD for 12 weeks
  Arms: Fesoterodine fumarate 8 mg (Double-Blind)
Drug: Placebo — Corresponding placebo tablets OD for 12 weeks
  Arms: Placebo (Double-Blind)
Drug: fesoterodine fumarate — 4mg tablets OD for 12 weeks
  Arms: Fesoterodine fumarate 4 mg (Double-Blind)

SUMMARY:
To evaluate the efficacy and safety of fesoterodine in comparison to placebo for overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Adult OAB patients who present with OAB symptoms, including micturitions >= 8 per day and urgency urinary incontinence >= 1 per day.

Exclusion Criteria:

* Patient has known hypersensitivity to the active substance (fesoterodine fumarate) or to peanut or soya or any of the excipients.
* Patient has a known neurological disease influencing bladder function.
* Patient has a complication of lower urinary tract pathology potentially responsible for urgency or incontinence, clinically relevant bladder outlet obstruction or pelvic organ prolapse.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 951 (Actual)
Dates: Start 2007-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (62):
- Hong Kong (2):
  - Pfizer Investigational Site, Kowloon
  - Pfizer Investigational Site, Shatin
- Japan (52):
  - Pfizer Investigational Site, Nagoya, Aichi-ken
  - Pfizer Investigational Site, Chuo-ku, Chiba-shi, Chiba
  - Pfizer Investigational Site, Eiheiji-cyo,yoshida-gun,, Fukui
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Koga-shi, Fukuoka
  - Pfizer Investigational Site, Minami-ku, Fukuoka-shi, Fukuoka
  - Pfizer Investigational Site, Nishiku, Fukuoka
  - Pfizer Investigational Site, Sawara-ku, Fukuoka
  - Pfizer Investigational Site, Amagasaki-shi, Hyōgo
  - Pfizer Investigational Site, Higashinada, Hyōgo
  - Pfizer Investigational Site, Nada-ku, Kobe-shi, Hyōgo
  - Pfizer Investigational Site, Suma-ku, Kobe-shi, Hyōgo
  - Pfizer Investigational Site, Takaraduka-city, Hyōgo
  - Pfizer Investigational Site, Aira-gun, Aira-chou,, Kagoshima-ken
  - Pfizer Investigational Site, Isogo-ku, Yokohama-shi, Kanagawa
  - Pfizer Investigational Site, Kawasakishi, Kanagawa
  - Pfizer Investigational Site, Sagamihara-shi, Kanagawa
  - Pfizer Investigational Site, Tama-ku, Kawasaki-shi, Kanagawa
  - Pfizer Investigational Site, Kochi, Kochi
  - Pfizer Investigational Site, Kumamoto, Kumamoto
  - Pfizer Investigational Site, Tamana-shi, Kumamoto
  - Pfizer Investigational Site, Matsumoto-shi, Nagano
  - Pfizer Investigational Site, Matumoto-Shi, Nagano
  - Pfizer Investigational Site, Hunaki-cho, Ibaraki-shi, Osaka
  - Pfizer Investigational Site, Kita-ku, Osaka-shi, Osaka
  - Pfizer Investigational Site, Kosobe-cho, Takatsuki-shi, Osaka
  - Pfizer Investigational Site, Minami-ku, Sakai-shi, Osaka
  - Pfizer Investigational Site, Nishinari-ku, Osaka
  - Pfizer Investigational Site, Osaka, Osaka
  - Pfizer Investigational Site, Suita-shi,, Osaka
  - Pfizer Investigational Site, Suita-shi, Osaka
  - Pfizer Investigational Site, Toyonaka, Osaka
  - Pfizer Investigational Site, Yodogawa-Ku, Osaka
  - Pfizer Investigational Site, Saitama-shi, Saitama
  - Pfizer Investigational Site, Satte-shi, Saitama
  - Pfizer Investigational Site, Wakou-shi, Saitama
  - Pfizer Investigational Site, Gotenbashi, Shizuoka
  - Pfizer Investigational Site, Susono, Shizuoka
  - Pfizer Investigational Site, Bunkyo-ku, Tokyo
  - Pfizer Investigational Site, Chofu-shi, Tokyo
  - Pfizer Investigational Site, Chuo-ku, Tokyo
  - Pfizer Investigational Site, Fucyushi, Tokyo
  - Pfizer Investigational Site, Koto-ku, Tokyo
  - Pfizer Investigational Site, Nakano-ku, Tokyo
  - Pfizer Investigational Site, Nishi-Tokyo-shi, Tokyo
  - Pfizer Investigational Site, Setagaya-ku, Tokyo
  - Pfizer Investigational Site, Setgaya-ku, Tokyo
  - Pfizer Investigational Site, Shibuya-ku, Tokyo
  - Pfizer Investigational Site, Shinjuku-ku, Tokyo
  - Pfizer Investigational Site, Suginami-ku, Tokyo
  - Pfizer Investigational Site, Sumida-ku, Tokyo
  - Pfizer Investigational Site, Chuou-shi, Yamanashi
- South Korea (3):
  - Pfizer Investigational Site, Cheonan-si, Chungcheongnam-do
  - Pfizer Investigational Site, Pusan
  - Pfizer Investigational Site, Seoul
- Taiwan (5):
  - Pfizer Investigational Site, Chiayi Country
  - Pfizer Investigational Site, Hualien City
  - Pfizer Investigational Site, Koahsiung
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Taipei

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221005&StudyName=Dose-Finding%20Study%20To%20Evaluate%20The%20Efficacy%2C%20Tolerability%20And%20Safety%20Of%20Fesoterodine%20In%20Comparison%20To%20Placebo%20For%20Overactive%20Bladder.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible subjects who underwent screening were enrolled into the run-in period at visit 1 and received single-blind placebo for 2 weeks. At Visit 2, Only subjects with overactive bladder who met the criteria were randomized to one of three treatment arms (fesoterodine 4 mg, fesoterodine 8 mg or placebo) in a 1:1:1 ratio.
Groups:
- Placebo: Subjects were treated with placebo once daily for 12 weeks.
- Fesoterodine 4 mg: Subjects were treated with Fesoterodine 4 mg/day for 12 weeks.
- Fesoterodine 8 mg: Subjects were treated with Fesoterodine 8 mg/day for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Fesoterodine 4 mg | Fesoterodine 8 mg
Started | 318 | 320 | 313
Completed | 285 | 286 | 281
Not Completed | 33 | 34 | 32
Not completed — Adverse Event | 11 | 14 | 14
Not completed — Lack of Efficacy | 5 | 3 | 2
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 10 | 9 | 10
Not completed — Protocol Violation | 4 | 3 | 4
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Meet Withdrawal Criterion | 0 | 1 | 1
Not completed — Adverse Event Occured Before Treatment | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Fesoterodine 4 mg | Fesoterodine 8 mg | Total
Number analyzed (Participants) | 318 | 320 | 313 | 951
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 227 | 217 | 196 | 640
  >=65 years | 91 | 103 | 117 | 311
Age Continuous [Mean (Standard Deviation); unit: years] | 56.7 (13.5) | 57.2 (14.2) | 58.8 (13.4) | 57.6 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 251 | 251 | 255 | 757
  Male | 67 | 69 | 58 | 194

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Number of Urgency Urinary Incontinence (UUI) Episodes Per 24 Hours at Week 12.
Description: Number of urgency urinary incontinence episodes was measured by the 3-day micturition diary completed for 3 consecutive days during the 7 days prior to each visit.
  Urgency urinary incontinence is the complaint of involuntary leakage accompanied by or immediately preceded by urgency. Urgency is the complaint of a sudden compelling desire to pass urine which is difficult to defer.
  Change: mean at Week 12 minus mean at Baseline.
Time Frame: Baseline to Week 12
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (95% Confidence Interval); unit: UUI Episodes
Arm/Group | Placebo | Fesoterodine 4 mg | Fesoterodine 8 mg
Number analyzed (Participants) | 309 | 314 | 306
UUI Episodes | -1.01 [-1.31 to -0.71] | -1.35 [-1.65 to -1.05] | -1.40 [-1.70 to -1.09]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 4 mg; The significance level was 0.05 (2-sided); Test type: Superiority or Other; p = 0.002, ANCOVA — The closed testing procedure was used in order to control the probability of a type 1 error; Analysis of covariance model with the treatment group, region as fixed effects and baseline values as a covariate was used; Mean Difference (Final Values) = -0.34, 95% CI [-0.56 to -0.13]
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine 8 mg; The significance level was 0.05 (2-sided); Test type: Superiority or Other; p < 0.001, ANCOVA — The closed testing procedure was used in order to control the probability of a type 1 error; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.39, 95% CI [-0.60 to -0.17]

2. Secondary Outcome: Change From Baseline in Mean Number of Urgency Urinary Incontinence (UUI) Episodes Per 24 Hours at Weeks 2, 4, 8, and 12.
Description: Number of urgency urinary incontinence (UUI) episodes was measured by the 3-day micturition diary completed for 3 consecutive days during the 7 days prior to each visit.
  Urgency urinary incontinence is the complaint of involuntary leakage accompanied by or immediately preceded by urgency. Urgency is the complaint of a sudden compelling desire to pass urine which is difficult to defer.
  Change: mean at each visit minus mean at Baseline.
Time Frame: Baseline to Weeks 2, 4, 8, and 12
Population: Full analysis set. No imputation was used for missing data.
Measure: Mean (Standard Deviation); unit: UUI Episodes
Arm/Group | Placebo | Fesoterodine 4 mg | Fesoterodine 8 mg
Number analyzed (Participants) | 309 | 314 | 306
UUI Episodes
  Week 2 (n=308, 314, 305) | -0.79 (1.465) | -1.10 (1.681) | -1.12 (1.736)
  Week 4 (n=301, 303, 296) | -1.15 (1.532) | -1.48 (1.688) | -1.49 (1.643)
  Week 8 (n=289, 289, 287) | -1.45 (1.518) | -1.61 (1.680) | -1.65 (1.690)
  Week 12 (n=284, 284, 281) | -1.49 (1.717) | -1.76 (1.618) | -1.87 (1.814)

3. Secondary Outcome: Change From Baseline in Mean Number of Micturitions Per 24 Hours at Week 12.
Description: Number of micturitions was measured by the 3-day micturition diary completed for 3 consecutive days during the 7 days prior to each visit.
  Change: mean at Week 12 minus mean at Baseline.
Time Frame: Baseline to Week 12
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (95% Confidence Interval); unit: Micturitions
Arm/Group | Placebo | Fesoterodine 4 mg | Fesoterodine 8 mg
Number analyzed (Participants) | 309 | 314 | 306
Micturitions | -0.59 [-1.08 to -0.10] | -1.15 [-1.64 to -0.67] | -1.25 [-1.75 to -0.76]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 4 mg; The significance level was 0.05 (2-sided); Test type: Superiority or Other; p = 0.002, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.56, 95% CI [-0.91 to -0.22]
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine 8 mg; The significance level was 0.05 (2-sided); Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.66, 95% CI [-1.01 to -0.32]

4. Secondary Outcome: Change From Baseline in Mean Number of Micturitions Per 24 Hours at Weeks 2, 4, 8, and 12.
Description: Number of micturitions was measured by the 3-day micturition diary completed for 3 consecutive days during the 7 days prior to each visit.
  Change: mean at each visit minus mean at Baseline.
Time Frame: Baseline to Weeks 2, 4, 8, and 12
Population: Full analysis set. No imputation was used for missing data.
Measure: Mean (Standard Deviation); unit: Micturitions
Arm/Group | Placebo | Fesoterodine 4 mg | Fesoterodine 8 mg
Number analyzed (Participants) | 309 | 314 | 306
Micturitions
  Week 2 (n=308, 314, 305) | -0.47 (1.786) | -0.94 (1.987) | -1.06 (2.076)
  Week 4 (n=301, 303, 296) | -0.85 (1.960) | -1.33 (2.146) | -1.60 (2.246)
  Week 8 (n=289, 289, 287) | -1.36 (2.215) | -1.81 (2.277) | -2.15 (2.402)
  Week 12 (n=284, 284, 281) | -1.36 (2.415) | -2.13 (2.214) | -2.17 (2.515)

5. Secondary Outcome: Change From Baseline in Mean Number of Urgency Episodes Per 24 Hours at Week 12.
Description: Number of urgency episodes was measured by the 3-day micturition diary completed for 3 consecutive days during the 7 days prior to each visit.
  Urgency is the complaint of a sudden compelling desire to pass urine which is difficult to defer.
  Change: mean at Week 12 minus mean at Baseline.
Time Frame: Baseline to Week 12
Population: Full analysis set. Last observation carried forward.
Measure: Least Squares Mean (95% Confidence Interval); unit: Urgency Episodes
Arm/Group | Placebo | Fesoterodine 4 mg | Fesoterodine 8 mg
Number analyzed (Participants) | 309 | 314 | 306
Urgency Episodes | -1.00 [-1.60 to -0.40] | -1.65 [-2.25 to -1.05] | -1.66 [-2.27 to -1.05]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 4 mg; The significance level was 0.05 (2-sided); Test type: Superiority or Other; p = 0.003, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.65, 95% CI [-1.07 to -0.22]
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine 8 mg; The significance level was 0.05 (2-sided); Test type: Superiority or Other; p = 0.002, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.66, 95% CI [-1.09 to -0.23]

6. Secondary Outcome: Change From Baseline in Mean Number of Urgency Episodes Per 24 Hours at Weeks 2, 4, 8, and 12.
Description: Number of urgency episodes was measured by the 3-day micturition diary completed for 3 consecutive days during the 7 days prior to each visit.
  Urgency is the complaint of a sudden compelling desire to pass urine which is difficult to defer.
  Change: mean at each visit minus mean at Baseline.
Time Frame: Baseline to Weeks 2, 4, 8, and 12
Population: Full analysis set. No imputation was used for missing data.
Measure: Mean (Standard Deviation); unit: Urgency Episodes
Arm/Group | Placebo | Fesoterodine 4 mg | Fesoterodine 8 mg
Number analyzed (Participants) | 309 | 314 | 306
Urgency Episodes
  Week 2 (n=308, 314, 305) | -0.79 (2.640) | -1.37 (2.722) | -1.59 (2.816)
  Week 4 (n=301, 303, 296) | -1.60 (2.780) | -2.16 (2.906) | -2.16 (3.065)
  Week 8 (n=289, 289, 287) | -2.34 (2.835) | -2.50 (3.080) | -2.71 (3.139)
  Week 12 (n=284, 284, 281) | -2.37 (2.975) | -2.89 (2.838) | -3.05 (3.462)

7. Secondary Outcome: Change From Baseline in Mean Number of Incontinence Episodes Per 24 Hours at Week 12.
Description: Number of incontinence episodes was measured by the 3-day micturition diary completed for 3 consecutive days during the 7 days prior to each visit.
  Incontinence is the complaint of any involuntary leakage of urine.
  Change: mean at Week 12 minus mean at Baseline.
Time Frame: Baseline to Week 12
Population: Full analysis set. Last observation carried forward
Measure: Least Squares Mean (95% Confidence Interval); unit: Incontinence Episodes
Arm/Group | Placebo | Fesoterodine 4 mg | Fesoterodine 8 mg
Number analyzed (Participants) | 309 | 314 | 306
Incontinence Episodes | -0.88 [-1.22 to -0.54] | -1.27 [-1.61 to -0.93] | -1.15 [-1.50 to -0.80]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 4 mg; The significance level was 0.05 (2-sided); Test type: Superiority or Other; p = 0.002, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.39, 95% CI [-0.63 to -0.14]
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine 8 mg; The significance level was 0.05 (2-sided); Test type: Superiority or Other; p = 0.030, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.27, 95% CI [-0.52 to -0.03]

8. Secondary Outcome: Change From Baseline in Mean Number of Incontinence Episodes Per 24 Hours at Weeks 2, 4, 8, and 12.
Description: Number of incontinence episodes was measured by the 3-day micturition diary completed for 3 consecutive days during the 7 days prior to each visit.
  Incontinence is the complaint of any involuntary leakage of urine.
  Change: mean at each visit minus mean at Baseline.
Time Frame: Baseline to Weeks 2, 4, 8, and 12
Population: Full analysis set. No imputation was used for missing data.
Measure: Mean (Standard Deviation); unit: Incontinence Episodes
Arm/Group | Placebo | Fesoterodine 4 mg | Fesoterodine 8 mg
Number analyzed (Participants) | 309 | 314 | 306
Incontinence Episodes
  Week 2 (n=308, 314, 305) | -0.80 (1.573) | -1.11 (1.725) | -1.06 (1.887)
  Week 4 (n=301, 303, 296) | -1.22 (1.598) | -1.61 (1.755) | -1.50 (1.707)
  Week 8 (n=289, 289, 287) | -1.56 (1.727) | -1.76 (1.795) | -1.73 (1.760)
  Week 12 (n=284, 284, 281) | -1.59 (1.869) | -1.97 (1.843) | -1.86 (2.000)

9. Secondary Outcome: Change From Baseline in Mean Number of Night-Time Micturitions Per 24 Hours at Week 12.
Description: Number of Night-Time Micturitions was measured by the 3-day micturition diary completed for 3 consecutive days during the 7 days prior to each visit.
  Change: mean at Week 12 minus mean at Baseline.
Time Frame: Baseline to Week 12
Population: Among the full analysis set, participants who had mean number of night-time micturitions per 24 hours of greater than 0 at baseline .
  Last observation carried forward.
Measure: Least Squares Mean (95% Confidence Interval); unit: Night-Time Micturitions
Arm/Group | Placebo | Fesoterodine 4 mg | Fesoterodine 8 mg
Number analyzed (Participants) | 243 | 256 | 257
Night-Time Micturitions | -0.18 [-0.41 to 0.06] | -0.21 [-0.44 to 0.02] | -0.29 [-0.52 to -0.05]
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine 4 mg; The significance level was 0.05 (2-sided); Test type: Superiority or Other; p = 0.624, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.04, 95% CI [-0.18 to 0.11]
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine 8 mg; The significance level was 0.05 (2-sided); Test type: Superiority or Other; p = 0.129, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.11, 95% CI [-0.26 to 0.03]

10. Secondary Outcome: Change From Baseline in Mean Number of Night-Time Micturitions Per 24 Hours at Weeks 2, 4, 8, and 12.
Description: Number of Night-Time Micturitions was measured by the 3-day micturition diary completed for 3 consecutive days during the 7 days prior to each visit.
  Change: mean at each visit minus mean at Baseline.
Time Frame: Baseline to Weeks 2, 4, 8, and 12
Population: Participants who had mean number of night-time micturitions per 24 hours of greater than 0 at baseline within the full analysis set.
  No imputation was used for missing data.
Measure: Mean (Standard Deviation); unit: Night-Time Micturitions
Arm/Group | Placebo | Fesoterodine 4 mg | Fesoterodine 8 mg
Number analyzed (Participants) | 243 | 256 | 257
Night-Time Micturitions
  Week 2 (n=242, 256, 256) | -0.25 (0.696) | -0.24 (0.796) | -0.34 (0.809)
  Week 4 (n=236, 246, 248) | -0.30 (0.835) | -0.30 (0.830) | -0.46 (0.780)
  Week 8 (n=224, 232, 241) | -0.41 (0.820) | -0.45 (0.815) | -0.58 (0.903)
  Week 12 (n=220, 229, 236) | -0.44 (0.945) | -0.48 (0.882) | -0.63 (0.945)

11. Secondary Outcome: Change From Baseline in Mean Voided Volume Per Micturition at Week 12.
Description: Voided volume per micturition was measured by the 3-day micturition diary completed for 3 consecutive days during the 7 days prior to each visit.
  Voided volume was recorded during any 1 day of 3-day diary period through the first micturition of the next day.
  Change: mean at Week 12 minus mean at Baseline.
Time Frame: Baseline to Week 12
Population: Full analysis set. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | Fesoterodine 4 mg | Fesoterodine 8 mg
Number analyzed (Participants) | 309 | 314 | 306
mL | 13.07 (46.207) | 22.80 (47.590) | 32.77 (52.893)

12. Secondary Outcome: Change From Baseline in Mean Voided Volume Per Micturition at Weeks 2, 4, 8, and 12.
Description: Voided volume per micturition was measured by the 3-day micturition diary completed for 3 consecutive days during the 7 days prior to each visit.
  Change: mean at each visit minus mean at Baseline.
Time Frame: Baseline to Weeks 2, 4, 8, and 12
Population: Full analysis set. No imputation was used for missing data.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | Fesoterodine 4 mg | Fesoterodine 8 mg
Number analyzed (Participants) | 309 | 314 | 306
mL
  Week 2 (n=308, 314, 304) | 5.06 (37.875) | 13.63 (35.350) | 21.52 (42.946)
  Week 4 (n=301, 303, 296) | 9.23 (43.639) | 21.62 (44.623) | 27.41 (45.803)
  Week 8 (n=289, 289, 287) | 10.75 (45.628) | 22.05 (44.949) | 30.94 (51.258)
  Week 12 (n=284, 284, 281) | 13.28 (46.317) | 24.52 (48.620) | 33.40 (53.379)

13. Secondary Outcome: Change From Baseline in Each Domain Scores of King's Health Questionnaire (KHQ).
Description: King's Health Questionnaire(KHQ) is used to assess the impact of bladder problems on quality of life. The each domain score was calculated valued and ranged from 0 to 100, where 0=best outcome/response and 100=worst outcome/response.
  Change: mean at Week 12 minus mean at Baseline.
Time Frame: Baseline to Week12
Population: Full analysis set. No imputation was used for missing data.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo | Fesoterodine 4 mg | Fesoterodine 8 mg
Number analyzed (Participants) | 285 | 283 | 283
score on scale
  General Health Perceptions (n=285, 283, 283) | -7.02 (22.573) | -9.36 (25.190) | -6.10 (25.272)
  Impact on Life (n=285, 283, 283) | -22.46 (28.018) | -27.33 (29.960) | -25.09 (32.172)
  Role Limitations (n=285, 283, 283) | -20.47 (27.730) | -27.92 (26.373) | -25.97 (28.590)
  Physical Limitations (n=285, 283, 283) | -18.65 (28.250) | -23.50 (28.807) | -25.97 (28.278)
  Social Limitations (n=285, 283, 283) | -14.44 (25.541) | -17.92 (24.029) | -18.53 (25.765)
  Personal Relationships (n=214, 210, 202) | -8.33 (21.773) | -16.11 (25.798) | -9.98 (24.335)
  Emotions (n=285, 283, 283) | -18.01 (26.365) | -24.70 (27.192) | -24.89 (27.310)
  Sleep/Energy (n=285, 283, 283) | -12.51 (24.967) | -19.08 (23.800) | -18.02 (25.287)
  Incontinence Severity Measures (n=285, 283, 283) | -13.75 (20.763) | -17.67 (21.038) | -18.59 (21.814)

14. Secondary Outcome: Change From Baseline in Each Domain Scores of Overactive Bladder Questionnaire (OAB-q) at Week 12.
Description: The overactive bladder questionnaire (OAB-q) is used to assess the extent of participants who had been bothered by selected bladder symptoms and to assess the effect on their health-related quality of life (HRQL).
  The each domain score ranges from 0 to 100 is a calculated value, where 0=minimal symptom severity and 100=greatest symptom severity for Symptom Bother Score, and where 0=worst HRQL outcome/response and 100=best HRQL outcome/response for HRQL domains including total score of HROL domain.
  Change: mean at Week 12 minus mean at Baseline.
Time Frame: Baseline to Week 12
Population: Full analysis set. Half scale rule (domain scores were calculated if a respondent had answered at least half of the items in a multi-item scale. Missing items were then replaced by the mean of non-missing items in that scale, for that participant.)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo | Fesoterodine 4 mg | Fesoterodine 8 mg
Number analyzed (Participants) | 285 | 283 | 283
score on scale
  Symptom Bother Score | -18.25 (23.618) | -26.61 (22.592) | -26.35 (23.849)
  Total Score of HRQL domain | 12.88 (18.868) | 17.84 (17.880) | 17.29 (19.670)
  Coping Score of HRQL domain | 16.54 (23.633) | 21.01 (22.109) | 21.48 (25.336)
  Concern Score of HRQL domain | 13.25 (21.182) | 20.05 (20.526) | 19.10 (21.868)
  Sleep Score of HRQL domain | 12.03 (22.215) | 16.16 (21.886) | 15.35 (24.654)
  Social Score of HRQL domain | 7.37 (17.211) | 11.35 (16.504) | 9.98 (16.706)

15. Secondary Outcome: Change From Baseline for Patient Perception of Bladder Condition (PPBC) at Week 12.
Description: Patient Perception of Bladder Condition (PPBC) score is rated on a 6-point scale as follows:
  1. No problems at all
  2. Some very minor problems
  3. Some minor problems
  4. Some moderate problems
  5. Severe problems
  6. Many severe problems
  Change: mean at Week 12 minus mean at Baseline.
Time Frame: Baseline to Week 12
Population: Full analysis set. No imputation was used for missing data.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo | Fesoterodine 4 mg | Fesoterodine 8 mg
Number analyzed (Participants) | 285 | 283 | 283
score on scale | -1.57 (1.236) | -1.83 (1.157) | -1.76 (1.182)

16. Secondary Outcome: The Number of Patients With "Severe Problems, Score 5" or "Many Severe Problems, Score 6" in Patient Perception of Bladder Condition (PPBC) at Week 12.
Description: Patient Perception of Bladder Condition (PPBC) score is rated on a 6-point scale as follows:
  1. No problems at all
  2. Some very minor problems
  3. Some minor problems
  4. Some moderate problems
  5. Severe problems
  6. Many severe problems
Time Frame: Baseline to Week 12
Population: Full analysis set. No imputation was used for missing data
Measure: Number; unit: participants
Arm/Group | Placebo | Fesoterodine 4 mg | Fesoterodine 8 mg
Number analyzed (Participants) | 285 | 283 | 283
participants
  Baseline | 82 | 97 | 83
  Week 12 | 28 | 12 | 19

ADVERSE EVENTS:
Arm/Group | Placebo | Fesoterodine 4 mg | Fesoterodine 8 mg
Serious Adverse Events (participants affected / at risk) | 5/318 | 3/320 | 0/313
Other Adverse Events (participants affected / at risk) | 68/318 | 138/320 | 185/313
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=318) | Fesoterodine 4 mg (N=320) | Fesoterodine 8 mg (N=313)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abscess (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=318) | Fesoterodine 4 mg (N=320) | Fesoterodine 8 mg (N=313)
Constipation (Gastrointestinal disorders) | 15 | 17 | 33
Cystitis (Infections and infestations) | 4 | 12 | 7
Diarrhoea (Gastrointestinal disorders) | 2 | 7 | 3
Dizziness (Nervous system disorders) | 1 | 7 | 2
Dry mouth (Gastrointestinal disorders) | 31 | 93 | 158
Dysuria (Renal and urinary disorders) | 0 | 2 | 14
Headache (Nervous system disorders) | 5 | 10 | 4
Nasopharyngitis (Infections and infestations) | 21 | 19 | 22
Residual urine (Renal and urinary disorders) | 5 | 7 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.